CLINICAL TRIAL: NCT05268536
Title: Comparison of the Effects of Core Stabilization and Resistance Exercises on Physical Fitness and Dance Performance in Latin Dancers
Brief Title: Comparison of the Effects of Core Stabilization and Resistance Exercises in Latin Dancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rüstem Mustafaoğlu, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-74555795-050.01.04-255256
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Dance
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resistance exercise (Active Comparator): Participants will perform Squat walking with resistance band, Butt blaster, Mussel with resistance band, Hip extension with resistance band, and Ankle dorsiflexion exercises with resistance band. All the participants will perform exercise for 6 weeks, 2 days a week for approximately 30-45 (including warm-up and cool-down).
  Interventions: Other: resistance exercise
- core stabilization exercise (Active Comparator): Patients will perform Plank, Bird dog, Double leg lifts, Prone cobra, Oblique twists exercises under the supervision of experienced Physiotherapist. All the participants will perform exercise for 6 weeks, 2 days a week for approximately 30-45 (including warm-up and cool-down).
  Interventions: Other: core stabilization exercise

INTERVENTIONS:
Other: core stabilization exercise — Patients will perform Plank, Bird dog, Double leg lifts, Prone cobra, Oblique twists exercises under the supervision of experienced Physiotherapist. All the participants will perform exercise for 6 weeks, 2 days a week for approximately 30-45 (including warm-up and cool-down).
  Arms: core stabilization exercise
Other: resistance exercise — resistance exercise
  Arms: resistance exercise

SUMMARY:
With our study, we aim to contribute to the literature by determining the effects of core stabilization and resistance exercise applications on muscle strength, endurance, balance, flexibility and performance in latin dancers. It is also aimed to raise awareness of the necessity of an exercise program in order to improve physical fitness parameters in addition to dance training in dancers. Considering the physiological demands of dance and dancer, it is necessary to develop a dance-specific approach by blending physical condition and art. Our study aims to contribute in this context.

DETAILED DESCRIPTION:
Within the scope of our study, the voluntary participation of 36 Latin dancers was planned. Dancers will be randomly divided into two groups, core stabilization exercises in one group and resistance exercises in the other group. An evaluation form developed by the researchers will be used as a data collection tool in the research. Before starting the study, a form containing demographic data (gender, age, height, weight, educational status) and medical history (chronic illness, previous injury, eating disorder) of the participants will be filled. Before starting the training, sit and stand test will be applied to evaluate the lower extremity muscle strength to evaluate the physical fitness parameters of the dancers, the plank test to evaluate the endurance, the Y balance test to evaluate the balance, the sit and reach test to evaluate the flexibility and the squat jump test to evaluate the performance. After the evaluation process, an exercise program for 6 weeks, 2 days a week and approximately 30-45 minutes (including warm-up and cool-down) will be applied for both groups. Core exercises will be applied to the 1st group, and resistance exercises will be applied to the 2nd group. Progress during the program will be achieved by increasing the intensity of the exercises. After 6 weeks of work, physical fitness parameters and performance will be evaluated again.

ELIGIBILITY:
Inclusion Criteria:

* • Being 18 years or older

  * Volunteering to participate in the study
  * Being actively attending latin dance lessons

Exclusion Criteria:

* • Being under the age of 18

  * Presence of upper or lower extremity musculoskeletal injuries or any cardiovascular, metabolic, neurological or pulmonary complications in the last 3 months
  * Being involved in any physiotherapy program in the last 3 months
  * Involvement in any exercise program other than dance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
sit to stand test | two weeks
  Within 30 seconds after the command is given, the participant repeats the full standing position from the fully seated position as quickly as possible. How many repetitions of sitting and standing are recorded during a 30-second period
plank test | two weeks
  The tester records in seconds how long the participant stayed in this position
Y balance test | two weeks
  There is an angle of 135 degrees between the rear strips and the front strip, and 45 degrees between the rear stripes. While trying to balance on one foot, the participant reaches out with the other foot in three different directions as far as possible. The specific test order is right anterior, left anterior, right posteromedial, left posteromedial, right posterolateral, and left posterolateral. The test manager records the participant's reach in centimeter to calculate the YBT composite distance.
sit and reach test | two weeks
  While sitting with the legs in a straight position, the person is asked to reach forward as far as possible without bending their knees, with their feet on a fixed object, with their hands on the coffee table, and wait for 2 seconds. In this position, the distance between the fingers and the object on which the foot rests is measured. Values before the object surface are recorded as negative, after values as positive, in centimeters
squat jump test | two weeks
  For a successful jump attempt, the participant must maintain the landing position for at least 2 seconds with her hands at waist level after the jump.

CONTACTS AND LOCATIONS:
Overall Officials: Rüstem Mustafaoğlu, PhD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No